CLINICAL TRIAL: NCT05057611
Title: Hemodynamic Phenotype-Based, Capillary Refill Time-Targeted Resuscitation In Early Septic Shock: The ANDROMEDA-SHOCK-2 Randomized Clinical Trial (A2)
Brief Title: Hemodynamic Phenotype and Capillary Refill Time-targeted Resuscitation Strategy
Acronym: A2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Fundacion Clinica Valle del Lili (Other); Hospital do Coracao (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021_02
Record Dates: First submitted 2021-09-06; First posted 2021-09-27 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (UC) (Active Comparator): - Patients allocated to the usual care group will be managed by the clinical staff according to usual practice at their sites including decisions about hemodynamic and perfusion monitoring, and all treatments, but should follow general recommendations of the Surviving Sepsis Campaign to avoid extremes of clinical practice. This includes basic hemodynamic targets such as a MAP >65 mmHg, HR (heart rate) <120 beats per minute (BPM), arterial oxygen saturation (SaO2) >94%, Hb > 7 gr/dl, and the use of NE as the first vasopressor and crystalloids as the fluid of choice.
  Interventions: Other: Usual care (UC)
- Capillary-refill time and phenotyping group (Experimental): Patients w/normal baseline CRT will be periodically monitored. Patients with abnormal CRT and septic shock will be categorized according to pulse pressure (PP). If <40 mmHg, will go to fluid responsiveness (FR) assessment. FR (-) patients will undergo cardiac echo to rule out significant dysfunction. Fluid boluses will be administered in 30 min intervals and repeated as needed if CRT is still abnormal. Patients with PP ≥40 mmHg will proceed according to diastolic pressure (DAP). If ≥50 mmHg will move to FR assessment. If <50 mmHg NE will be increased for MAP >65 mmHg and DAP ≥50 mmHg w/CRT assessed 1 h after. NE will be increased in 0.1 mcg/k/m increments up to 0.5 mcg/k/m.
  If CRT is normal, patients will proceed to periodic monitoring. Patients with persistent abnormal CRT or that reached NE safety limit will proceed directly to echo.
  Patients that correct CRT with first tier interventions will not be subjected to obligatory echo but will just proceed to periodic monitoring.
  Interventions: Other: CRT-targeted strategy associated with a clinical hemodynamic phenotyping to personalize initial resuscitation in septic shock patients

INTERVENTIONS:
Other: CRT-targeted strategy associated with a clinical hemodynamic phenotyping to personalize initial resuscitation in septic shock patients — A combination of combine a CRT-targeted strategy with a clinical hemodynamic phenotyping that may aid to personalize initial resuscitation with potential additional fluid-sparing effects.
  Arms: Capillary-refill time and phenotyping group
Other: Usual care (UC) — - Patients allocated to the UC group will be managed by the clinical staff according to usual practice at their sites including decisions about hemodynamic and perfusion monitoring, and all treatments, but should follow general recommendations of the Surviving Sepsis Campaign to avoid extremes of clinical practice. This includes basic hemodynamic targets such as a MAP >65 mmHg, heart rate (HR) <120 beats per minute (BPM), arterial oxygen saturation (SaO2) >94%, Hb > 7 gr/dl, and the use of NE as the first vasopressor and crystalloids as the fluid of choice.
  Arms: Usual Care Group (UC)

SUMMARY:
Septic shock is associated with a high mortality risk. Fluid overload occurs when fluids are administered to fluid unresponsive patients, but also when inappropriate resuscitation goals are pursued. Alongside, evidence confirms that abnormal peripheral perfusion after resuscitation is associated with increased morbidity and mortality. Targeted resuscitation associates with lower mortality, less organ dysfunction, and less intensity of treatment. Over-resuscitation may contribute to a worse outcome.

Many patients remain hypovolemic after initial resuscitation. Others present very low diastolic arterial pressures (DAP) reflecting profound vasoplegia and may benefit from early norepinephrine (NE) instead of fluids. Administering fluids in this setting could increase the risk of fluid overload. In addition, relevant myocardial dysfunction is present in a significant number of patients. Pulse pressure (PP) and DAP evaluation may help clinicians to individualize initial management sparing unnecessary fluid loading.

Objective: To test if a CRT-targeted resuscitation based on clinical hemodynamic phenotyping can improve a hierarchical clinical outcome - mortality, time to cessation of vital support, and length of hospital stay, all within 28 days - in septic shock patients as compared to usual care.

A2 is a multicenter randomized controlled trial (RCT) comparing a CRT-targeted, hemodynamics-based resuscitation strategy with usual care in patients with early septic shock during a 6 h intervention period. A sample size of 1500 patients was calculated to detect a 6% absolute reduction in mortality in the CRT group, and the win-ratio method will be used to test the superiority in the hierarchical outcomes mentioned above.

The combination of a CRT-targeted strategy with a clinical hemodynamic phenotyping may aid to personalize initial resuscitation with potential additional fluid-sparing effects. To categorize patients at baseline according to PP may conduct patients with low PP (<40mmHg) to fluid responsiveness (FR) assessment and eventually fluid boluses, while patients with normal PP will be treated according to DAP, adjusting NE when to avoid further fluids loading in patients who normalize CRT.

Fluid resuscitation will be focused on FR+ hypoperfused patients to prevent harmful fluid administration in FR- patients.

DETAILED DESCRIPTION:
I. Introduction Septic shock is associated with a high mortality risk related to progressive tissue hypoperfusion. However, despite extensive research on the best monitoring and resuscitation strategies, many uncertainties remain. Over-resuscitation, particularly when inducing fluid overload, might contribute to a worse outcome. Fluid overload more likely occurs when fluids are administered to fluid unresponsive patients, but also when inappropriate resuscitation goals are pursued, or a "one-size-fits-all" strategy is followed.

From a hemodynamic point of view, several pathogenic mechanisms determine a progressive circulatory dysfunction. While loss of vascular tone and relative hypovolemia predominate in early phases, more complex mechanisms such as endothelial and microcirculatory dysfunction, progressive vasoplegia, and myocardial dysfunction may be involved later. In effect, from a clinical point of view, many patients despite been fluid loaded in pre-intensive care unit (ICU) settings, are still evidently hypovolemic and benefit from further administration of fluid boluses. Others, however, present very low diastolic arterial pressures (DAP) reflecting profound vasoplegia, and recent data suggest that these patients may benefit from early norepinephrine (NE) instead of fluids on the contrary, administering fluids may fail to correct vascular tone and increase the risk of fluid overload. In addition, a recent echocardiography-based study confirmed that a relevant myocardial dysfunction is present in a significant number of patients and that several cardiovascular phenotypes with a potentially different therapeutic approach may be recognized. Despite research efforts, no universally applicable clinical phenotyping method for septic shock patients has been translated to usual practice. This is particularly problematic since echocardiography is not immediately available in the majority of centers worldwide, and therefore initial decisions on fluid resuscitation are usually based on clinical grounds and tend to follow the "one-size-fits-all" principle, leading to the risk of fluid overload.

II. ANDROMEDA-SHOCK Study The excellent prognosis associated with CRT recovery, its rapid-response time to fluid loading, its relative simplicity, its availability in resource-limited settings, and its capacity to change in parallel with perfusion of physiologically relevant territories such as the hepatosplanchnic region, constitute strong reasons to consider CRT as the target for fluid resuscitation in septic shock patients.

ANDROMEDA-SHOCK was a multicenter, randomized controlled trial comparing CRT- versus lactate-targeted resuscitation in patients with early septic shock. The main outcome was 28-day mortality, and secondary outcomes included organ dysfunction and treatment intensity. The hypothesis was that targeting CRT would lead to decreased mortality and organ dysfunction due to less fluid administration and treatment intensity.

CRT-targeted resuscitation was associated with lower mortality (34.9% vs. 43.4%), beneficial effects on organ dysfunction, and less intensity of treatment. The superiority of this strategy was also supported by a subsequent Bayesian analysis. The key novelty of A2 is to combine a CRT-targeted strategy with a clinical hemodynamic phenotyping that may aid to personalize initial resuscitation with potential additional fluid-sparing effects.

III. Rationale for ANDROMEDA-SHOCK-2 intervention strategy. There are four relevant actions that may increase the efficacy of A2 intervention strategy to decrease mortality and organ dysfunction due to potential fluid-sparing effects or at least by promoting a more rational septic shock resuscitation.

1. Use of CRT as a target A key aspect of ANDROMEDA-SHOCK was a more rational approach to fluid resuscitation based on selecting a more appropriate target such as CRT. In fact, almost a 25% of patients assigned to the CRT arm had a normal CRT at baseline, and thus received no further fluid resuscitation. This fact is per se fluid sparing. In addition, a significant number of patients corrected CRT at 2h with initial fluid boluses. This rapid response of CRT to flow-increasing maneuvers makes CRT particularly suitable as a target. In addition, a recent clinical-physiological study suggested that normalization of CRT was associated to resolution of profound tissue hypoperfusion as assessed by hypoxia surrogates, and regional/sublingual microcirculatory variables. For these reasons and other considerations described elsewhere, a CRT-targeted resuscitation will be applied as the intervention arm of A2.
2. Clinical hemodynamic phenotyping Hypotension assessed by mean arterial pressure (MAP) is the hallmark of sepsis-related acute circulatory dysfunction, and since duration of hypotension is related to morbidity and mortality, current guidelines recommend fluids and vasopressors administered in a stepwise fashion to increase MAP levels to >65 mmHg to ensure minimal organ perfusion pressure. This "MAP-driven strategy" has probably led to an unwanted side-effect, a reductionist approach to clinical hemodynamic monitoring where among numerous variables provided by the blood pressure signal, only MAP is considered for decision-making at the bedside. Moreover, this standardized resuscitation strategy is debatable since septic shock patients are highly heterogeneous. For example, a recent report showed that 30% of septic shock patients admitted to ICU were already fluid unresponsive, and others have suggested that early start of NE instead of fluids could be associated with better outcomes in predominantly vasoplegic patients.

   Pulse pressure (PP) as a surrogate of stroke volume. In normal conditions, DAP is mainly determined by vascular tone and it remains nearly constant from the ascending aorta to the peripheral vessels. Thus, detection of low DAP at peripheral vessels should reflect systemic vasodilation as long as the aortic valve is competent. However, DAP is not considered for septic shock definition, and with few exceptions, its relationship with clinical outcomes has not been widely described. Nevertheless, evaluation of the loss of vascular tone through the severity of diastolic hypotension could have profound implications on therapeutic decisions since there are not robust clues to rapidly predict when hypotension will be sustainably corrected with fluid loading. Thus, rapid assessment of severity of vasodilation could influence therapeutic decisions such as the early introduction of NE, which theoretically may avoid unnecessary fluid administration while promptly restoring tissue perfusion. A low DAP (<50 mmHg) may impair myocardial perfusion of the left ventricle (LV), especially in the case of tachycardia where diastolic time is limited.
3. Systematic and repeated assessment of fluid responsiveness.

   Fluid administration is the first line therapy to reverse sepsis-induced tissue hypoperfusion. For this purpose, fluids are administered either as fluid loading at the emergency department, or later as fluid challenges during advanced ICU-based resuscitation. However, as any other drug, fluids have a narrow therapeutic index. Insufficient fluid resuscitation may lead to progressive tissue hypoperfusion and organ dysfunction, while excess fluids could induce detrimental fluid overload.

   Fluid responsiveness (FR) is a physiological cardiovascular condition where an increase in preload induced by a fluid bolus leads to an increase in cardiac output (CO) by more than 10-15%. In non-fluid responsive (FR-) patients, fluid administration does not significantly increase CO and may contribute to congestion and fluid overload. The rationale to assess FR is then to try to optimize fluid resuscitation in critically ill patients by focusing fluid boluses in FR+ hypoperfused patients and by preventing harmful fluid administration in FR- patients.

   Multiple tests have been described to assess FR at the bedside. They allow to determine the position of the patient's heart on its systolic function curve and are based upon changes in cardiac output or stroke volume resulting from various changes in preload conditions, induced by heart-lung interactions, postural maneuvers or by the infusion of small amounts of fluids. By applying the appropriate tests, FR can be assessed in a wide variety of clinical settings. However, despite their relative simplicity, lack of cost, and side effects, the use of FR tests has not completely permeated into routine clinical practice. One of the contributing factors is that even under the optimal conditions of their use, their sensitivity and specificity is not perfect, and all have significant limitations. This may be linked to the unreliability of the test, but also to the lack of precision of the measurement method used to estimate its effects.

   In A2, FR assessment will be performed systematically in every patient with abnormal CRT randomized to the intervention arm and presenting a low PP. FR assessment will be repeated after every fluid bolus (500 ml of crystalloids in 30 minutes) to decide on further fluid administration if CRT target was not achieved. A FR- status or a safety issue may command to move to other steps of the intervention algorithm.
4. Selective Critical Care Echocardiography

IV. Usual Care group Recruited centers for A2 should exhibit a historical mortality for septic shock of <40%. Patients allocated to the control (usual care) group will be managed by the clinical staff according to usual practice at their sites including decisions about hemodynamic and perfusion monitoring, and all treatments, but should follow general recommendations of the Surviving Sepsis Campaign to avoid extremes of clinical practice.

All data regarding insertion of invasive monitoring devices, intravenous-fluid resuscitation, vasoactive support, mechanical ventilation, and other supportive therapies will be collected by the study coordinator or monitors. Lead investigators at a site will not serve as the bedside treating physician for patients in the usual-care group.fluid administration in FR- patients.

V. Physiological substudies Several substudies will be performed in all or part of the participating centers including venous congestion substudy (VExUS), sublingual microcirculation substudy, and renal doppler resistive index substudies. These substudies are highly relevant since they will compare the impact of A2 intervention strategy on effective organ perfusion microcirculatory flow, and venous congestion, thus determining if this resuscitative strategy is associated with a more harmonic resuscitation as expressed by a "perfusion without congestion" result.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients (≥ 18 years) with septic shock according to Sepsis-3 consensus conference (septic shock defined as suspected or confirmed infection, plus hyperlactatemia and NE requirements due to persistent hypotension, after a fluid load of at least 1000 mL in one hour)

Exclusion Criteria:

* More than 4 hours since septic shock diagnosis,
* Anticipated surgery or acute hemodialysis procedure to start during the 6h intervention period
* Active bleeding,
* Do not resuscitate status,
* Child B-C Cirrhosis
* Underlying disease process with a life expectancy < 90 days and/or the attending clinician deems aggressive resuscitation unsuitable
* Refractory shock (high risk of death within 24h)
* Pregnancy
* Concomitant severe acute respiratory distress syndrome.
* Patients in whom CRT cannot be accurately assessed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
A composite of all cause 28-days mortality plus time to cessation of vital support and length of hospital stay | 28 days
  A hierarchical composite of all cause mortality within 28 days, time to cessation of vital support (truncated at 28 days) and length of hospital stay (truncated at 28 days).

SECONDARY OUTCOMES:
All-cause mortality within 28 days | 28 days
  All-cause mortality within 28 days
Vital support free days | 28 days
  The number of calendar days between randomization and 28 days that the patient is alive and with no requirement of cardiovascular, respiratory and renal support. Patients who die within 28 days will have zero days counted for this variable, irrespective of vital support status.
  Resolution of cardiovascular failure implies complete stopping of vasopressor support for at least 24 consecutive hours. Resolution of respiratory failure implies extubation / liberation from mechanical ventilation for at least 48 hours. Resolution of renal failure implies liberation of renal replacement therapy for at least 72 hours in those receiving continuous replacement modalities and at least 5 days for those receiving intermittent ones.
Length of hospital stay | 28 days
  Number of days remaining hospitalized (from randomization up to hospital discharge), truncated at day 28.

OTHER OUTCOMES:
Length of ICU stay | 28 days
  Number of days remaining in ICU (from randomization up to ICU discharge). Re-admission to ICU during follow-up period will be accounted for the original ICU length of stay only if occurred within the next week of ICU discharge and by a cause related with the original admission.
Time to cessation of vasopressor support | 28 days
  The number of hours between randomization and complete stopping of vasopressor support (defined as its complete interruption for at least 24 consecutive hours), within 28 days from randomization.
Time to cessation of mechanical ventilation | 28 days
  The number of calendar days between intubation / start of mechanical ventilation and extubation / liberation from mechanical ventilation (maintained for at least 48 hours) within 28 days from randomization.
Time to cessation of renal replacement therapy | 28 days
  The number of calendar days between start of renal replacement therapy and complete liberation from renal replacement therapy (at least 48 hours for continuous replacement modalities and 5 days for intermittent ones) within 28 days from randomization.
Vasopressor support-free days | 28 days
  The number of calendar days without vasopressor support from randomization up to day 28. Cessation of vasopressor support implies its complete interruption for at least 24 consecutive hours.
Mechanical ventilation-free days | 28 days
  The number of calendar days without mechanical ventilation support from randomization up to day 28. Cessation of mechanical ventilation support implies its complete interruption for at least 48 consecutive hours.
  Re-start of mechanical ventilation during follow-up period will be accounted for the original mechanical ventilation-free days only if this occurs within the next week of ICU discharge and by a cause related with the original admission.
Renal replacement therapy-free days | 28 days
  The number of calendar days without renal replacement therapy from randomization up to day 28. Cessation of renal replacement therapy implies its complete interruption for at least 72 hours in those receiving continuous replacement modalities and at least 5 days for those receiving intermittent ones.
  Re-start of renal replacement therapy during follow-up period will be accounted for the original renal replacement-free days only if this occurs within the next week of ICU discharge and by a cause related with the original admission.
Variation in Sequential Organ Failure Assessment (SOFA) score | 7 days
  The Sequential Organ Failure Assessment (SOFA) is used to track a patient's status during the stay in the ICU to determine the extent of organ dysfunction. Its values ranges from 0 to 24. Higher SOFA scores associate with a worse outcome.
  The SOFA score will be calculated upon the maximum values observed on the day of enrollment and then, at days 2, 3, 4, 5 and 7 (or until patient discharge or death, if this happened before day-7), using clinically available data. If an individual organ dysfunction value is not available (i.e., cardiovascular, respiratory, renal, etc.), it will be assumed to be zero unless previous value was abnormal (in which case it would be considered the same organ score). Neurological score under sedation/invasive mechanical ventilation will be computed as that observed just before sedation/intubation.
Variation of creatinine-based KDIGO stage | 7 days
  Renal function assessed according to "Kidney Disease: Improving Global Outcomes (KDIGO) staging system from randomization through day 7 to assess for "de novo" or "worsening" acute kidney injury. Patients under chronic renal replacement therapy will not meet this end-point
Volume of resuscitation fluids | 72 hours
  The volume of fluids administered with resuscitative intention up to 72 hours from randomization.
Net fluid balance | 72 hours
  The volume of cumulated fluids during the first 72 hours from randomization.
Evolvement of capillary refill time (CRT) | 72 hours
  Evolvement of CRT within the first 72 hours after randomization.
Evolvement of lactate levels | 72 hours
  Evolvement of arterial lactate levels within the first 72 hours after randomization.
Evolvement of central venous pressure | 72 hours
  Evolvement of Central venous pressure within the first 72 hours after randomization.
Evolvement of central venous oxygen saturation | 72 hours
  Evolvement of central venous oxygen saturation within the first 72 hours after randomization.
Evolvement of central venous to arterial carbon dioxide difference | 72 hours
  Evolvement of central venous to arterial carbon dioxide difference within the first 72 hours after randomization.
All-cause mortality within 90 days | 90 days
  All-cause mortality within 90 days
Length of hospital stay | 90 days
  Number of days remaining hospitalized (from randomization up to hospital discharge), truncated at day 90.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Hernandez, MD, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] ANDROMEDA-SHOCK-2 Investigators for the ANDROMEDA Research Network, Spanish Society of Anesthesiology, Reanimation and Pain Therapy (SEDAR), and Latin American Intensive Care Network (LIVEN); Hernandez G, Ospina-Tascon GA, Kattan E, Ibarra-Estrada M, Ramasco F, Orozco N, Ramos K, Aldana JL, Ferri G, Hamzaoui O, De Backer D, Teboul JL, Vieillard-Baron A, Petri Damiani L, Garcia-Gallardo GA, Morales S, Carmona Garcia P, Mendez R, Hernandez-Gilsoul T, Perez-Nieto OR, Olea Vielba C, Ramos S, Dominguez D, Bruna M, David S, Wendel-Garcia PD, Galiana-Ivars M, Myatra SN, Messina A, Cecconi M, Pozo M, Amthauer M, Higuera E, Al Duhalib Z, Rico-Feijoo J, Ferrer-Gomez C, Perez-Carbonell A, Martinez-Castro S, Redondo Calvo FJ, Vives M, Sanchez HF, Bilbao I, Fernandez P, Al-Fares A, Benitez-Cano A, Gonzalez C, Reyes LF, Rodriguez-Guillen JH, Cristino AV, Pendino JC, Ortiz G, Alonso-Gonzalez MC, Murias G, Aguirre-Avalos G, Hernandez L, Calderon Barajas ZA, Zarragoikoetxea I, Monnet X, Goury A, Mendonca Dos Santos T, Vallecilla L, Martins de Lima L, Sady E, Alegria L, Ostermann M, Bakker J, Biasi Cavalcanti A. Personalized Hemodynamic Resuscitation Targeting Capillary Refill Time in Early Septic Shock: The ANDROMEDA-SHOCK-2 Randomized Clinical Trial. JAMA. 2025 Dec 9;334(22):1988-1999. doi: 10.1001/jama.2025.20402. PMID 41159835
- [Derived] Prager R, Argaiz E, Pratte M, Rola P, Arntfield R, Beaubien-Souligny W, Denault AY, Haycock K, Miralles Aguiar F, Bakker J, Ospina-Tascon G, Orozco N, Rochwerg B, Lewis K, Quazi I, Kattan E, Hernandez G, Basmaji J. Doppler identified venous congestion in septic shock: protocol for an international, multi-centre prospective cohort study (Andromeda-VEXUS). BMJ Open. 2023 Jul 24;13(7):e074843. doi: 10.1136/bmjopen-2023-074843. PMID 37487682
- [Derived] Kattan E, Bakker J, Estenssoro E, Ospina-Tascon GA, Cavalcanti AB, Backer D, Vieillard-Baron A, Teboul JL, Castro R, Hernandez G. Hemodynamic phenotype-based, capillary refill time-targeted resuscitation in early septic shock: The ANDROMEDA-SHOCK-2 Randomized Clinical Trial study protocol. Rev Bras Ter Intensiva. 2022 Jan-Mar;34(1):96-106. doi: 10.5935/0103-507X.20220004-pt. PMID 35766659